CLINICAL TRIAL: NCT07168200
Title: A Randomized, Controlled, Double-blind, Multicenter Phase III Clinical Study of Adebrelimab Combined With Concurrent Chemoradiotherapy Versus Placebo Combined With Concurrent Chemoradiotherapy for the Treatment of Locally Advanced Cervical Cancer
Brief Title: A Phase III Clinical Study of Adebrelimab Combined With Concurrent Chemoradiotherapy Versus Placebo Combined With Concurrent Chemoradiotherapy for the Treatment of Locally Advanced Cervical Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Shengdi Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR-1316-305
Record Dates: First submitted 2025-09-04; First posted 2025-09-11 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Advanced Cervical Cancer
MeSH Terms: interventions — Cisplatin; Carboplatin; Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHR-1316 Group (Experimental)
  Interventions: Drug: SHR-1316 Injection; Drug: Cisplatin Injection; Drug: Carboplatin Injection; Drug: Paclitaxel Injection
- SHR-1316 Placebo Group (Placebo Comparator)
  Interventions: Drug: Cisplatin Injection; Drug: Carboplatin Injection; Drug: Paclitaxel Injection; Drug: SHR-1316 Placebo Injection

INTERVENTIONS:
Drug: SHR-1316 Injection — SHR-1316 injection.
  Arms: SHR-1316 Group
Drug: Cisplatin Injection — Cisplatin injection.
Drug: Carboplatin Injection — Carboplatin injection.
Drug: Paclitaxel Injection — Paclitaxel injection.
Drug: SHR-1316 Placebo Injection — SHR-1316 placebo injection.
  Arms: SHR-1316 Placebo Group

SUMMARY:
This study aims to evaluate the efficacy of Adebrelimab plus concurrent chemoradiotherapy compared with placebo plus concurrent chemoradiotherapy for the treatment of locally advanced cervical cancer by evaluating progression-free survival (PFS).

ELIGIBILITY:
Inclusion Criteria:

1. Participate in the study voluntarily, sign the informed consent form.
2. Subjects were able to provide primary or metastatic cancer samples.
3. At least one measurable lesion.
4. Expected survival > 3 months.
5. ECOG 0 ~ 1.
6. With adequate organ functions.

Exclusion Criteria:

1. Pathologically or radiologically confirmed presence of distant metastatic disease, including lymph nodes above the first lumbar vertebra (L1) (cephalad) or in the inguinal region.
2. Administering live vaccines within 4 weeks before enrollment or during planned study treatment.
3. Participants who received immunosuppressive therapy within 4 weeks before enrolment.
4. For participants who are receiving thrombolytic/anticoagulant therapy, prophylactic anticoagulant therapy is allowed.
5. Participants who have had other uncured malignant tumors in the past (within 5 years) or concurrently have had other uncured malignant tumors, excluding cured basal cell carcinoma of the skin and carcinoma in situ.
6. Known allergy to the investigational drug or any of its excipients; or severe allergic reaction to other monoclonal antibodies.
7. Pregnant or breastfeeding women.
8. According to the investigator's judgment, there are diseases or any other conditions that may seriously endanger the safety of the subjects, may confound the research results, or affect the subjects' ability to complete the study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 720 (Estimated)
Dates: Start 2025-10-17 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Up to approximately 36 months.

SECONDARY OUTCOMES:
Overall survival (OS) | Up to approximately 60 months.
  OS is the time interval from the start of treatment to death due to any reason or lost of follow-up.
3-year overall survival (OS) rate | Up to approximately 60 months.
  OS rate within 3 years.
2-year progression-free survival (PFS) | Up to approximately 24 months.
  PFS within 2 years.
Objective Response Rate (ORR) | Up to approximately 36 months.
Duration of response (DoR) | Up to approximately 60 months.
Local progression rate | Up to approximately 36 months.
Distant recurrence rate | Up to approximately 60 months.
The second disease progression assessed by the investigator | Up to approximately 60 months.
Adverse events (AEs) including incidence and grade correlation with study drugs | Up to approximately 60 months.
Rate of suspension and discontinuation due to an adverse event correlation with study drugs | Up to approximately 60 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided